CLINICAL TRIAL: NCT00391300
Title: Development of an Electrical Diagnostic for Melanoma and Other Cutaneous Malignancies
Brief Title: Bioelectric Field Imaging in Diagnosing Melanoma and Other Skin Cancers in Patients With Skin Lesions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: CDR0000616117; EVMS-BFI and Lesions
Record Dates: First submitted 2006-10-02; First posted 2006-10-23 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2008-10

CONDITIONS: Melanoma (Skin); Non-melanomatous Skin Cancer
Keywords: melanoma; basal cell carcinoma of the skin; squamous cell carcinoma of the skin
MeSH Terms: conditions — Melanoma; Carcinoma, Basal Cell | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: bioelectric field imaging
Procedure: biopsy
Procedure: histopathologic examination

SUMMARY:
RATIONALE: New diagnostic procedures, such as bioelectric field imaging, may help find and diagnose melanoma and other skin cancers. It may also be a less invasive way to check for skin cancer.

PURPOSE: This phase I trial is studying bioelectric field imaging in diagnosing melanoma and other skin cancers in patients with skin lesions.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if the hand-held Bioelectric Field Imager can be used to measure the electric field in skin of various body surfaces, including face, neck, shoulders, arms, hands, chest, back, legs, and feet, during the course of examination and treatment of patients with suspected malignant skin lesions.
* To determine if there is a significant difference between the lateral electric field strength near benign and malignant skin lesions in the same individual.

OUTLINE: Patients undergo scanning of their skin lesions and nearby healthy skin using the Bioelectric Field Imager (BFI). The lesions are then biopsied for histological diagnosis. Histological data from the biopsy is correlated with the electric field data from the BFI.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Suspected malignant skin lesion
* Seeking treatment for skin lesion at the VA Medical Center

PATIENT CHARACTERISTICS:

* Not pregnant
* No acute illness, including upper respiratory tract infection or flu that could result in fever
* No trauma to the skin lesion area
* No prisoners

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-04 (Estimated); Study Completion 2007-04 (Estimated)

PRIMARY OUTCOMES:
Use of Bioelectric Field Imager (BFI) in measuring the electric field in skin of various body surfaces
Use of BFI in detecting significant electric field differences between malignant and benign skin lesions

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette F. Hood, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- VA Hospital, Hampton, Virginia, United States